CLINICAL TRIAL: NCT00135278
Title: Cerebrospinal Fluid (CSF) Drainage and Cytokine Profiling in the Treatment of Acute Spinal Cord Injury (SCI) - A Pilot Study
Brief Title: Cerebrospinal Fluid (CSF) Drainage and Cytokine Profiling in the Treatment of Acute Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brian Kwon, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C04-0584; V05-0160
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injuries
Keywords: Neuroprotection; inflammation; cytokines; CSF
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSF Drainage (Other)
  Interventions: Procedure: CSF Drainage
- No CSF Drainage (Other)
  Interventions: Procedure: No CSF Drainage

INTERVENTIONS:
Procedure: CSF Drainage — See Detailed Description
  Arms: CSF Drainage
Procedure: No CSF Drainage — See Detailed Description
  Arms: No CSF Drainage

SUMMARY:
The overall purpose of this pilot study is to evaluate CSF drainage as a potential neuroprotective strategy after acute spinal cord injury (SCI).

DETAILED DESCRIPTION:
This pilot study will evaluate the safety and feasibility of a clinical trial protocol for cerebrospinal fluid (CSF) drainage as a potential treatment for patients with acute spinal cord injury. Specifically, the investigators will evaluate:

* patient eligibility and recruitment for such a study and how soon CSF drainage can be instituted in such patients;
* adverse events and safety of CSF drain insertion and drainage in the setting of acute spinal cord injury;
* neurologic recovery after injury; and
* cytokine expression within the CSF and blood after injury.

Following informed consent, patients with spinal cord injuries who agree to participate in the study will have a lumbar CSF drain placed and be randomized to either:

* CSF drainage to maintain a constant intrathecal pressure; or
* no CSF drainage.

Both groups will have CSF and blood sampled at pre-defined intervals in order to evaluate CSF cytokine expression after acute spinal cord injury. For comparison against the injured condition, CSF and blood from a normal group of uninjured individuals will be obtained. These individuals will be patients undergoing hip or knee surgery under a spinal anesthetic, where a small sample of CSF can be taken when their intrathecal space is accessed for the anesthesia.

Outcomes that will be measured in spinal cord injured patients include the eligibility and recruitment rate of patients, the time required to institute lumbar drainage, and adverse effects related to CSF drain insertion and CSF drainage. Neurologic function will be measured according to American Spinal Injury Association (ASIA) standards. Patient-reported quality of life and functional independence measurements will be evaluated. CSF and serum will be evaluated for the expression of inflammatory cytokines.

The results of this pilot study will provide feasibility and safety information that will be critical in the both the decision to pursue and in the planning of a larger prospective randomized clinical trial to formally assess the clinical efficacy of CSF drainage as a therapy for patients with acute spinal cord injury.

BACKGROUND INFORMATION/STUDY RATIONALE

Traumatic Spinal Cord Injuries - Epidemiology and Research Overview:

Few traumas to the human body are as suddenly and permanently devastating as spinal cord injuries. Unfortunately, it is most often young, highly productive, otherwise healthy adults who sustain such injuries, and thereafter suffer lifelong loss of movement, sensation, and bowel, bladder, and sexual function. In North America, over 10,000 people sustain a spinal cord injury each year, and currently there are estimated to be over 250,000 individuals living with chronic spinal cord paralysis (Sekhon and Fehlings, 2001). Important advances in medical, surgical, and rehabilitative treatments have improved the clinical care of spinal cord injured patients over the past few decades. Nevertheless, there are still no convincingly effective treatments currently available to improve the neurological status of these patients, and as such, their paralysis is currently an incurable condition.

This rather dismal neurologic prognosis has stimulated significant research efforts to understand the neurobiology of spinal cord injury and develop effective therapies for it. This international effort has tremendously increased our understanding of the neuropathology of spinal cord injury and has shed much insight into the acute and chronic pathophysiologic processes that inhibit neural regeneration and functional recovery (reviewed by Kwon et al., 2002). The large majority of research into spinal cord repair strategies can be conceptually divided into two streams:

* research on the acute pathophysiologic processes that occur immediately or soon after injury, with the aim of developing neuroprotective therapies that attenuate these processes to minimize secondary spinal cord damage; and
* research on the intrinsic and extrinsic impediments to axonal re-growth within the central nervous system, with the aim of developing axonal regeneration therapies that would promote axonal growth across the injured spinal cord and thus mediate recovery after spinal cord injury (Kwon et al., 2004a).

Pathophysiology of Traumatic Spinal Cord Injuries - The Role of Ischemia:

The majority of individuals who sustain spinal cord injuries do not suffer a complete transection of their spinal cords, even if they have functionally complete paralysis. Rather, while the initial "primary" mechanical impact interrupts axons at the site of injury and disrupts the local neuronal and glial cytoarchitecture, a proportion of the spinal cord (usually the outer rim) escapes intact. This spared tissue, however, is then subject to a complex cascade of acute pathophysiologic processes that cause further "secondary" damage. These interrelated processes include ionic homeostasis abnormalities, excitotoxicity, programmed cell death, tissue ischemia, and inflammation (Kwon et al., 2004b). Neuroprotective therapies aim to counteract these processes, thereby averting further secondary damage and maximizing the extent of spared cord tissue. Animal studies have demonstrated that significant neurologic function can be mediated by small amounts of spared cord tissue, and in this regard, even small neuroprotective effects might reap substantial functional benefits to patients.

Vascular disruption and local tissue ischemia have long been recognized as important aspects of secondary damage following acute traumatic spinal cord injury. Ischemia and resultant cellular energy failure is thought to contribute to the propagation of many other important pathophysiologic processes, and in this regard has been argued by some to be the most critical component of secondary damage (Amar and Levy, 1999). Mechanical disruption of the microvasculature causes petechial hemorrhage and intravascular thrombosis, which in combination with vasospasm of intact vessels and edema at the injury site can lead to profound local hypoperfusion and ischemia (Tator and Fehlings, 1991). This is primarily a microvascular phenomenon, with the larger caliber vessels such as the anterior spinal artery normally being spared (Koyanagi et al., 1993). Human post-mortem studies have demonstrated that vascular perfusion is substantially worse in the grey matter than in the white matter, which may be related to the disruption and/or thrombosis of the sulcal arterial network that centrifugally supplies much of the grey matter (Tator and Koyanagi, 1997). The high metabolic requirements of neurons make the grey matter exquisitely sensitive to ischemia injury, which can be compounded by the loss of autoregulatory mechanisms which normally maintain fairly constant microvascular hemodynamics within the spinal cord during systolic blood pressure fluctuations (Senter and Venes, 1979). The loss of autoregulation makes the cord vulnerable to further ischemic insult from systemic hypotension (Kobrine et al., 1975).

The Role of Ischemia in Non-Traumatic Spinal Cord Injury:

Up to this point, the discussion has focused on spinal cord injuries caused by blunt trauma and the role that ischemia plays in the secondary injury cascade. Ischemia alone, however, can also be the primary etiologic process behind paralysis in non-traumatic circumstances. Such is the case in patients undergoing thoracoabdominal aortic aneurysm (TAAA) repair. In these surgeries, the aorta is clamped and segmental vessels ligated, thus depriving the spinal cord of its blood supply to an extent that is influenced by the severity and location of the aneurysm and the duration of the vascular occlusion. The incidence of paralysis caused by this ischemic insult has been estimated between 3.8 to 17.6% (Crawford and Rubio, 1973), but has been reported to be as high as 28 to 41% after the repair of particular types of aneurysms (Crawford et al., 1986; Safi et al., 1996). As perioperative paraplegia is one of the most devastating complications of this surgery, a number of adjunctive treatments have been investigated as prophylactic or therapeutic interventions. These include generalized or local hypothermia, medications such as steroids, naloxone, barbiturates, papaverine, reattachment of intercostal arteries, and CSF drainage (Wan et al., 2001). In principle, these interventions aim to reduce spinal cord ischemia by either improving vascular perfusion (increasing cellular oxygen supply) or by reducing metabolic activity (decreasing cellular oxygen demand).

CSF Drainage as a Method for Preventing or Treating Spinal Cord Ischemia:

The drainage of CSF has emerged as an accepted intervention for reducing the risk of ischemic paralysis in patients undergoing thoracoabdominal aortic aneurysm repair. An important determinant of oxygen supply to the spinal cord is the spinal cord perfusion pressure (SCPP), defined as the gradient between mean distal aortic arterial pressure (MDAP) and CSF pressure (CSFP) (WADA et al., 2001). Conceptually, the drainage of CSF reduces CSF pressure and thus increases the perfusion pressure and oxygen delivery to the spinal cord. When cross clamping of the aorta occurs, the distal aortic pressure decreases and the gradient between arterial and CSF pressure narrows. Additionally, a significant increase in CSF pressure has been demonstrated to occur with aortic cross-clamping itself (WADA et al., 2001), which would serve to further reduce the spinal cord perfusion pressure. The reasons for this increase in CSF pressure with aortic cross-clamping are unclear, but may be related to changes in venous capacitance causing sequestration of venous blood within the dura and bony neural axis (Piano and Gewertz, 1990). Seminal animal experiments performed decades ago demonstrated that following descending aortic occlusion, a decrease of arterial pressure to or below that of CSF pressure (decreasing SCPP) almost universally resulted in paraplegia, while the drainage of CSF to reduce CSF pressure (and thus increase SCPP) was effective in preventing paraplegia. (MIYAMOTO et al., 1960; Oka and Miyamoto, 1987).

Since then, numerous clinical reports have described the use of CSF drainage in humans undergoing TAAA repair (reviewed by Ling, 2000 [Ling and Arellano, 2000]). Normal CSF pressure in humans has been documented to be approximately 13 to 15 mmHg (Drenger et al., 1997). Increased CSF pressures of 21 to 25 mm Hg have been demonstrated with aortic cross clamping (Drenger et al., 1997; WADA et al., 2001) . It has been advocated therefore to drain CSF in a controlled manner to maintain CSF pressure at approximately 10 mm Hg during TAAA repair (Carroccio et al., 2003). A prospective randomized controlled trial by Svensson et al. demonstrated a 12% (2 of 17) incidence of neurologic deficit in patients treated with CSF drainage compared to a 44% (7 of 16) incidence in the control group (p=0.0392) (Svensson et al., 1998). A more recent prospective randomized controlled trial of 145 patients by Coselli et al. demonstrated with an intent-to-treat analysis a significant reduction in paraplegia with CSF drainage to keep the CSF pressure around 10 mmHg (Coselli et al., 2002). Neurologic deficits occurred in 2 of 82 patients (2.7%) undergoing CSF drainage and 9 of 74 patients (12.2%) in the control group (p=0.026), representing an 80% reduction in relative risk. Both of these prospective randomized studies were terminated early at a planned interim analysis due to the significant benefit demonstrated by CSF drainage. Of note, complications related to the CSF drainage, such as headache, meningitis, or subdural hemorrhage were not observed in these studies.

These prospective randomized studies illustrate the potential efficacy of CSF drainage in preventing paraplegia when the spinal cord is subjected to ischemic insult. In addition to this, CSF drainage has been reported to be effective as a treatment in cases where the ischemic insult has already resulted in paraplegia. Such reports are obviously relevant to traumatic spinal cord injuries in which some ischemic damage would likely already be present by the time CSF drainage was instituted. Ackerman and Traynelis reported on the institution of CSF drainage in 6 patients who suffered ischemic paralysis, 5 of whom were between 12 and 40 hours post-TAAA repair (Ackerman and Traynelis, 2002). In four patients who had their CSF drainage started within 14 hours of the onset of their ischemic symptoms, significant neurologic recovery was achieved. In three of these patients, the neurologic recovery occurred immediately after the CSF catheter was inserted. In two patients who had their CSF drainage started 32 and 27 hours after the onset of symptoms, no neurologic recovery was observed. Safi et al. reported on the initiation of CSF drainage in 8 patients presenting with neurologic deficits 1 to 14 days after TAAA repair (Safi et al., 1997). They observed substantial neurologic recovery of at least 2 Frankel grades in all 8 patients. The interpretation of these results requires acknowledgement of the fact that other treatments such as steroids and vascular support were also instituted, but they do suggest that the principles of modulating spinal cord perfusion pressure with CSF drainage are still applicable in patients who have already suffered ischemic injury to the spinal cord.

The Inflammatory Reaction to Spinal Cord Injury and CSF Cytokines:

As stated earlier, secondary damage to the spinal cord after the initial mechanical impact is mediated by a number of pathophysiologic processes, including ionic homeostasis abnormalities, excitotoxicity, programmed cell death, tissue ischemia, and inflammation. The preceding discussion has focused on tissue ischemia and how this might be affected by CSF drainage. Inflammation appears to also play an important role in the pathophysiology of acute spinal cord injury, and has thus been the focus of increasing attention in recent years. The inflammatory response to spinal cord injury is mediated by cytokines that influence vascular permeability and regulate migration of inflammatory cells such as neutrophils and macrophages into the spinal cord (Kwon et al., 2004b). The list of cytokines thought to be relevant to the inflammatory response after spinal cord injury is long, and includes IL-1 , IL-1 , TNF , IL-6, IL-10, VEGF, and a variety of leukotrienes. (Mueller et al., 2003;Widenfalk et al., 2003; Mitsuhashi et al., 1994; Xu et al., 1990; Bartholdi and Schwab, 1997; Carmel et al., 2001; Hayashi et al., 2000; Pan et al., 2002; Wang et al., 1997) Recently, a study of the injured spinal cords of 11 patients who died shortly after their trauma demonstrated the presence of IL-1 , IL-6, and TNF positive cells within the spinal cord within 24 hours of injury. (Yang et al., 2004)

While some aspects of the inflammatory and immunologic response mediated by these cytokines may be beneficial after spinal cord injury, others may be detrimental. (Bethea, 2000) For example, after a contusion spinal cord injury, transgenic mice lacking the TNF receptor were found to have increased apoptosis, a larger area of secondary injury, and worse locomotor scores than wild-type mice. (Kim et al., 2001) Conversely, the systemic administration of IL-10 significantly reduced neuronal damage after an excitotoxic spinal cord injury. (Brewer et al., 1999) A more sophisticated understanding of these complex responses is obviously needed. Nevertheless, these animal studies demonstrate the proof of concept that the manipulation of these cytokine responses has the potential to influence outcome after spinal cord injury, and therefore, may represent the targets for neuroprotective intervention. The levels of expression for each cytokine appear to change over time and the temporal specificity of the expression likely also influences the inflammatory response.

Are CSF Cytokine Measurements Representative of the Events in the Cord?:

Without question, the most direct method of examining the cytokine response after spinal cord injury would be to obtain samples of the cord itself. While this has largely been the method by which such phenomena have been examined in animal models, it is obviously not possible in living human patients. The recent study by Yang et al. evaluated the spinal cord tissue from patients who had died, but did not sample the CSF to determine how closely the cord changes were reflected in the CSF space. In a rat spinal cord contusion injury model, Wang et al. demonstrated an increase in IL-1 in both the spinal cord tissue itself and in the CSF.(Wang et al., 1997) While the IL-10 concentration was much lower in the CSF than in the cord, the increase in IL-10 in the CSF after spinal cord injury paralleled the increase observed in the cord. These animal data suggest that cytokine analysis of the CSF can provide some meaningful data about what is happening within the cord.

There is, to our knowledge, only one human study that has examined cytokine levels within the CSF of patients after acute blunt spinal cord injury. This study examined levels of the eicosanoids, LTC4, TXB2, and 6-keto-PGF1 between 0 and 17 days post-injury, and then again at 6 months post-injury.(Nishisho et al., 1996) These authors found an increase in all three eicosanoids, and found that LTC4 levels correlated to some extent with injury severity. In a study of patients undergoing thoracoabdominal aortic aneurysm repair (possibly inducing ischemic insults to the spinal cord), Kunihara et al. demonstrated increased levels of IL-8 that were independent of serum levels, and in particular noted sustained IL-8 elevation in a patient who unfortunately became paraplegic after the operation.(Kunihara et al., 2001) In a study of CSF from adult patients with severe brain injury, Csuka et al demonstrated increases in IL-10 that were independent of serum IL-10 levels.(Csuka et al., 1999) While direct comparison with the spinal cord tissue is not possible in these human studies, they do suggest that CNS injury is associated with cytokine changes that can be detected in the CSF.

The involvement of cytokines in the inflammatory process and their presence in the CSF raises the potential for an additional benefit to CSF drainage which has not yet been explored in humans. Kunihara and colleagues demonstrated a significant increase in the pro-inflammatory cytokine interleukin-8 (IL-8) within the spinal cords of New Zealand white rabbits subjected to aortic cross-clamping (Kunihara et al., 2000). They went on to show that levels of IL-8 (in addition to other inflammatory cytokines such as IL-10 and IL-6) were significantly elevated in the CSF of human patients undergoing TAAA repair. Interestingly, a patient in this series who suffering ischemic paraplegia after the TAAA had the most dramatically increased and sustained levels of IL-8 within the CSF (Kunihara et al., 2001). It has been proposed by these authors and others that the drainage of such pro-inflammatory CSF cytokines away from the spinal cord may itself be neuroprotective (Kunihara et al., 2001; Tang et al., 1996; Svensson et al., 1998). This hypothesis, however, has not been further evaluated in traumatic or non-traumatic spinal cord injuries. As yet, it is unclear how much CSF would need to be drained in order to achieve an "effective" reduction in local cytokine concentration.

Summary:

In summary, the drainage of CSF has been shown in human clinical studies to be neuroprotective in the setting of ischemic injury to the spinal cord, both with respect to prevention and treatment. Given that ischemia is also a well recognized contributor to the secondary injury cascade following traumatic spinal cord injury, there is a cogent rationale for the evaluation of CSF drainage in this setting, acknowledging the desperate need for the development of effective treatments for such patients. To our knowledge, there have been no previously reported evaluations of CSF drainage in human patients who have suffered an acute traumatic spinal cord injury.

Also, given the enormous current worldwide interest in the inflammatory response to spinal cord injury, it is reasonable to conclude that promising experimental neuroprotective interventions will be forthcoming within the near future. If such strategies are to be moved from the animal models within the laboratory setting and into human patients, it would be extremely useful to characterize the inflammatory response in humans and compare it to available animal data. Such knowledge would not only be helpful in predicting which experimental therapies would be beneficial, but also would be helpful in the definition of parameters for monitoring the effectiveness of therapeutic interventions. In this regard, changes in cytokines/chemokines may become an additional outcome measure for the evaluation of therapeutic efficacy. Moreover, insights gained here may direct laboratory (animal) studies towards clinically relevant parameters.

ELIGIBILITY:
Inclusion Criteria:

Injured subjects:

* Complete or incomplete acute SCI between C0 and T11
* Admitted within 48 hours of injury
* Undergoing spinal decompressive surgery
* Undergoing lumbar puncture for spinal anesthetic or myelography
* Neurologically intact

Exclusion Criteria:

* Pre-existing neurodegenerative disorder
* Associated head or spine injury

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01-27 (Actual); Study Completion 2010-01-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and feasibility of CSF drainage as a potential treatment for patients with acute SCI

SECONDARY OUTCOMES:
To determine if CSF drainage will improve neurologic function after acute SCI
To evaluate the temporal pattern of expression of inflammatory cytokines within the CSF

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Brian Kwon, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Stukas S, Cooper J, Gill J, Fallah N, Skinnider MA, Belanger L, Ritchie L, Tsang A, Dong K, Streijger F, Street J, Paquette S, Ailon T, Dea N, Charest-Morin R, Fisher CG, Bailey CS, Dhall S, Mac-Thiong JM, Wilson JR, Christie S, Dvorak MF, Wellington CL, Kwon BK. Association of CSF and Serum Neurofilament Light and Glial Fibrillary Acidic Protein, Injury Severity, and Outcome in Spinal Cord Injury. Neurology. 2023 Mar 21;100(12):e1221-e1233. doi: 10.1212/WNL.0000000000206744. Epub 2023 Jan 4. PMID 36599698